CLINICAL TRIAL: NCT04842253
Title: High Flow Nasal Cannula (HFNC) Versus Standard Low Flow Nasal Cannula (LFNC) in Patients with Atrial Fibrillation Undergoing Radiofrequency Catheter Ablation (RFCA) Under Deep Desaturation.
Brief Title: HFNC Vs LFNC in Patients with AF Undergoing RFCA Under Deep Sedation.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to changes in logistics (indications Rf and attendance PFA), it has not been feasible to include the required number of participants in this study
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72859
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Deep Sedation; Oxygen Therapy; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High flow nasal cannula (Experimental): Participants in the high flow nasal cannula group will receive high flow nasal cannula oxygen during deep sedation.
  Interventions: Device: High flow nasal cannula
- Low flow nasal cannula (No Intervention): Participants in the current standard of care will receive low flow nasal cannula during deep sedation.

INTERVENTIONS:
Device: High flow nasal cannula — HFNC during deep sedation undergoing radiofrequency ablation for atrial fibrillation.
  Other Names: High flow nasal oxygen
  Arms: High flow nasal cannula

SUMMARY:
Oxygen supplementation through high flow nasal cannula (HFNC) may reduce the incidence of desaturation and hypoxemia during deep sedation at radiofrequency catheter ablation (RFCA procedures).This study is designed to test the hypothesis that the incidence of hypoxemia and desaturation in patients with atrial fibrillation undergoing RFCA under deep sedation, is less when using HFNC as compared to use of standard low flow nasal cannula (LFNC).

DETAILED DESCRIPTION:
Desaturation may occur in patients under deep sedation which results in an elevated risk for perioperative adverse events including hypoxemia (1-3). The incidence of hypoxemia was 168 per 1000 in a general procedural sedation and analgesia population (4). The clinical significance of transient episodes of hypoxemia remains debatable. However, many peri-operative incidents are often short-term and limited in nature, but a number of them are a predictor to a serious complication with a permanent injury (5).This study investigates if high flow nasal cannula (HFNC) as compared to low flow nasal cannula (LFNC) will result in a lower incidence of intra-procedural oxygen desaturation and hypoxemia in patients with atrial fibrillation undergoing deep sedation for radiofrequency catheter ablation (RFCA).

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing an elective RFCA for atrial fibrillation in the Maastricht UMC Cardiac Catheter Labs under deep sedation administered by a clinician anesthesiology

Exclusion Criteria:

* Age under 18 years
* Body Mass Index (BMI) > 32 kg/m²
* Diagnosed Sleep Apnoea Syndrome (SAS)
* Chronic Pulmonary Obstructive Disease (COPD) gold IV and COPD gold III with frequent or recent exacerbation
* Diagnosed pulmonary or cardiac condition requiring chronic oxygen therapy
* Complete nasal obstruction
* Active nose bleeding
* Untreated pneumothorax (pre- existing)
* Recent upper airway surgery
* Recent base of skull fracture
* Expected difficult airway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Hypoxemia event | The outcome variable will be measured during the patient's sedation (0-4 hours).
  The primary outcome measure will be the lowest measured blood oxygen level during the patient's sedation.

SECONDARY OUTCOMES:
Duration of hypoxemia event | The outcome variable will be measured during the patient's sedation (0-4 hours).
  The secondary outcome measure will be the duration of the lowest measured blood oxygen level during the patient's sedation.
Cross over from oxygen therapy | The outcome variable will be measured during the patient's sedation (0-4 hours).
  The secondary outcome measure will be cross over from oxygen therapy during sedation yes/no.
To measure the incidence of hypoxemia and desaturation (SpO2 under 90% for > 60 seconds). | The outcome variable will be measured during the patient's sedation (0-4 hours).
  The secondary outcome measure will be the incidence SpO2 under 90% for > 60 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Esther AC Bouman, Doctor, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht UMC, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share IPD is still undecided because we are not certain if we are going to share all collected IPD or all IPD that underlie results in a publication.

REFERENCES:
- [Background] Jirapinyo P, Thompson CC. Sedation Challenges: Obesity and Sleep Apnea. Gastrointest Endosc Clin N Am. 2016 Jul;26(3):527-37. doi: 10.1016/j.giec.2016.03.001. PMID 27372775
- [Background] Qadeer MA, Rocio Lopez A, Dumot JA, Vargo JJ. Risk factors for hypoxemia during ambulatory gastrointestinal endoscopy in ASA I-II patients. Dig Dis Sci. 2009 May;54(5):1035-40. doi: 10.1007/s10620-008-0452-2. Epub 2008 Nov 12. PMID 19003534
- [Background] Salukhe TV, Willems S, Drewitz I, Steven D, Hoffmann BA, Heitmann K, Rostock T. Propofol sedation administered by cardiologists without assisted ventilation for long cardiac interventions: an assessment of 1000 consecutive patients undergoing atrial fibrillation ablation. Europace. 2012 Mar;14(3):325-30. doi: 10.1093/europace/eur328. Epub 2011 Oct 23. PMID 22024600
- [Background] Conway A, Sutherland J. Depth of anaesthesia monitoring during procedural sedation and analgesia: A systematic review and meta-analysis. Int J Nurs Stud. 2016 Nov;63:201-212. doi: 10.1016/j.ijnurstu.2016.05.004. Epub 2016 May 25. PMID 27236824
- [Background] Koers L, Eberl S, Cappon A, Bouwman A, Schlack W, Hermanides J, Preckel B. Safety of moderate-to-deep sedation performed by sedation practitioners: A national prospective observational study. Eur J Anaesthesiol. 2018 Sep;35(9):659-666. doi: 10.1097/EJA.0000000000000835. PMID 29847362
- [Background] Sago T, Watanabe K, Kawabata K, Shiiba S, Maki K, Watanabe S. A Nasal High-Flow System Prevents Upper Airway Obstruction and Hypoxia in Pediatric Dental Patients Under Intravenous Sedation. J Oral Maxillofac Surg. 2021 Mar;79(3):539-545. doi: 10.1016/j.joms.2020.10.018. Epub 2020 Oct 16. PMID 33176129
- [Derived] Homberg MC, Bouman EA, Linz D, van Kuijk SMJ, Joosten BA, Buhre WF. High-flow nasal cannula versus standard low-flow nasal cannula during deep sedation in patients undergoing radiofrequency atrial fibrillation catheter ablation: a single-centre randomised controlled trial. Trials. 2022 May 9;23(1):378. doi: 10.1186/s13063-022-06362-1. PMID 35534903